CLINICAL TRIAL: NCT06580522
Title: The Effect of the Position Given to the Child After Weaning from Noninvasive Mechanical Ventilation on Physiological Symptoms
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Acibadem University (Other)
Collaborators: Istanbul University - Cerrahpasa (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Supportive Care
Other Study IDs: 2023/30
Record Dates: First submitted 2024-08-02; First posted 2024-08-30 (Actual); Last update posted 2024-08-30 (Actual); Status verified 2024-08

CONDITIONS: Prone Position; Supine Position; Child
MeSH Terms: conditions — Deception

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Prone Position Group (Experimental): Children in this group were given the prone position after weaning from noninvasive mechanical ventilation and its effect on the physiologic symptoms of the children was examined.
  Interventions: Other: Prone Position Group
- Supine Position Group (Experimental): Supine position group children were given supine position after weaning from noninvasive mechanical ventilation and the effects on physiologic symptoms were examined.
  Interventions: Other: Supine Position Group

INTERVENTIONS:
Other: Prone Position Group — After the children in the prone position group were weaned from noninvasive mechanical ventilation according and started to breathe spontaneously, they were prone positioned and monitored for 120 minutes (2 hours) every 20 minutes (0.min, 20.min, 40.min, 60.min, 80.min, 100.min, 120.min) with a head-monitor for peak heart rate, oxygen saturation, respiratory rate and blood pressure.
  Arms: Prone Position Group
Other: Supine Position Group — After the children in the supine position group were weaned from noninvasive mechanical ventilation according and started to breathe spontaneously, they were supine positioned and monitored for 120 minutes (2 hours) every 20 minutes (0.min, 20.min, 40.min, 60.min, 80.min, 100.min, 120.min) with a head-monitor for peak heart rate, oxygen saturation, respiratory rate and blood pressure.
  Arms: Supine Position Group

SUMMARY:
The aim of this clinical trial was to investigate the effect of the position given to children after weaning from noninvasive mechanical ventilation on the physiological symptoms (heart rate, oxygen saturation, respiratory rate and blood pressure) of children aged six months to six years in the Pediatric Intensive Care Unit.

ELIGIBILITY:
Inclusion Criteria:

* Between 6 months and 6 years of age
* Being monitored for respiratory diseases
* Weaning from noninvasive mechanical ventilation during the research process
* Body temperature within the normal range (36 centigrade-37,5 centigrade)
* Verbal and written consent to participate in the study given by their parents

Exclusion Criteria:

* Congenital anomaly
* Surgical intervention that prevents supine/prone positioning
* Development of pneumothorax during research
* Hypoxia during the research

Ages: 6 Months to 6 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 40 (Actual)
Dates: Start 2023-03-01 (Actual); Primary Completion 2024-07-26 (Actual); Study Completion 2024-07-26 (Actual)

PRIMARY OUTCOMES:
Pulse changes in children after weaning from noninvasive mechanical ventilation | 120 minutes after weaning from noninvasive mechanical ventilation
  Changes in the pulse rate of children will be measured and recorded at 20 minute intervals for 120 minutes after the position given to the children after weaning from noninvasive mechanical ventilation. The changes in the pulse rate values of the children between the age groups in the study in terms of minutes/pulse rate and the difference values between them according to minutes will be examined.

OTHER OUTCOMES:
Oxygen saturation changes in children after weaning from noninvasive mechanical ventilation | 120 minutes after weaning from noninvasive mechanical ventilation
  Changes in oxygen saturation values of children will be measured and recorded at 20 minute intervals for 120 minutes after the position given to children after weaning from noninvasive mechanical ventilation. The changes in % of oxygen saturation values of children between the age groups in the study and the difference values between them according to minutes will be analyzed.
Respiratory rate changes in children after weaning from noninvasive mechanical ventilation | 120 minutes after weaning from noninvasive mechanical ventilation
  Changes in respiratory rate values of children will be measured and recorded at 20 minute intervals for 120 minutes after the position given to children after weaning from noninvasive mechanical ventilation. The changes in the respiratory rate values of the children between the age groups in the study in minutes/respiratory rate and the difference values between them according to minutes will be examined.
Blood pressure changes in children after weaning from noninvasive mechanical ventilation | 120 minutes after weaning from noninvasive mechanical ventilation
  Changes in blood pressure values of children will be measured and recorded at 20 minute intervals for 120 minutes after the position given to children after weaning from noninvasive mechanical ventilation. The changes in the blood pressure values of the children in mm/Hg between the age groups in the study and the difference values between them according to minutes will be examined.

CONTACTS AND LOCATIONS:
Overall Officials: Duygu Gözen, Prof.Dr., Study Director — Koç Üniversitesi
Locations (1):
- Istanbul University Cerrahpasa Medical Faculty Hospital, Istanbul, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No